CLINICAL TRIAL: NCT00902174
Title: A 24-week Randomized Placebo-controlled, Double-blind Multi-center Clinical Trial Evaluating the Efficacy and Safety of Oral QTI571 as an add-on Therapy in the Treatment of Severe Pulmonary Arterial Hypertension: Imatinib in Pulmonary Arterial Hypertension, a Randomized, Efficacy Study (IMPRES)
Brief Title: Imatinib (QTI571) in Pulmonary Arterial Hypertension
Acronym: IMPRES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQTI571A2301
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2013-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Imatinib; 6MWD; Borg scale; Pulmonary hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- imatinib mesylate (Experimental): Imatinib mesylate (QTI571) 200 mg once daily for two weeks, increased to 400 mg once daily if well tolerated. If 400 mg dose was not well tolerated, a down titration to 200 mg once daily was permitted.
  Interventions: Drug: imatinib mesylate
- Placebo (Placebo Comparator): Placebo to imatinib mesylate taken once daily. Participants receiving placebo were allowed to receive already approved PAH treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: imatinib mesylate — Two or 4 imatinib mesylate (QTI571) 100 mg film coated tablets once daily.
  Arms: imatinib mesylate
Drug: Placebo — Placebo to imatinib 100 mg film coated tablets
  Arms: Placebo

SUMMARY:
A multinational, multicenter, double blind, placebo-controlled study evaluating the efficacy and safety of imatinib as an add-on therapy in the treatment of patients with severe pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Key Inclusion criteria

* Male or female patients ≥18 years of age with a current diagnosis of pulmonary arterial hypertension (PAH) according to the Dana Point 2008 Meeting: World Health Organization (WHO) Diagnostic Group I, idiopathic or heritable (familial or sporadic) PAH, PAH associated with collagen vascular disease including systemic sclerosis, rheumatoid arthritis, mixed connective tissue diseases, and overlap syndrome. PAH following one year repair of congenital heart defect [Atrial Septal Defect (ASD), Ventricular Septal Defect (VSD) or Posterior Descending Artery (PDA)], or PAH associated with diet therapies or other drugs
* A Pulmonary Vascular Resistance (PVR) ≥ 800 dynes.sec.cm-5 (as assessed by Right Heart Catheterization (RHC) at screening or in the 3 months preceding the screening visit) despite treatment with two or more specific PAH therapies, including Endothelin Receptor Antagonists (ERAs), phosphodiesterase 5 inhibitors (PDE5), or subcutaneous, inhaled, intravenous or oral prostacyclin analogues for ≥ 3 months. Background therapy doses were to be stable for ≥ 30 days except for warfarin and prostacyclin analogues ( ≥ 30 days but doses could vary even within the month before enrollment).
* World Health Organization functional Class II-IV. For WHO Functional Class IV, one of the 2 or more specific PAH therapies were to be an inhaled, subcutaneous, intravenous or oral prostacyclin analogue, unless the subject showed intolerance of prostacyclin analogues.
* 6MWD ≥ 150 meters and ≤ 450 meters at screening. Distances of two consecutive 6MWTs were to be within 15% of one another.

Key Exclusion criteria

* With a pulmonary capillary wedge pressure > 15 mm Hg to rule out PAH secondary to left ventricular dysfunction.
* With a diagnosis of pulmonary artery or vein stenosis
* Left ventricular ejection fraction (LVEF) < 45%
* With Disseminated Intravascular Coagulation (DIC)
* With evidence of major bleeding or intracranial hemorrhage
* With a history of elevated intracranial pressure
* With a history of latent bleeding risk such as diabetic retinopathy, gastrointestinal bleeding due to gastric or duodenal ulcers, or colitis ulcerosa
* With a QTcF > 450 msec for males and > 470 msec for females at screening and baseline in the absence of right bundle branch block.
* With a history of ventricular tachycardia, ventricular fibrillation or ventricular flutter
* With a history of Torsades de Pointes
* With a history of long QT syndrome
* Having undergone atrial septostomy in the 3 months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (90):
- United States (28):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Miami Beach, Florida
  - Novartis Investigative Site, Weston, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Minneola, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Austria (2):
  - Novartis investigative site, Innsbruck
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Canada (7):
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, Edmonton
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Ottawa
  - Novartis investigative site, Toronto
  - Novartis Investigative Site, Vancouver
- Novartis Investigative Site, Clamart, France
- Germany (13):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis investigative site, Löwenstein
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensberg
  - Novartis Investigative Site, Würzberg
- Italy (4):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Roma
- Japan (6):
  - Novartis Investigative Site, Bunkyō City
  - Novartis Investigative Site, Hamamatsu
  - Novartis Investigative Site, Mitaka
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Sendai
  - Novartis Investigative Site, Suita
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Seoul, South Korea
- Spain (12):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Caceras
  - Novartis Investigative Site, Las Palmas de Gran Canarias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis investigative site, San Cristóbal de La Laguna
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Seville
  - Novartis investigative site, Valencia
  - Novartis Investigative Site, Valladolid
- Sweden (4):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - University Hospital Basel, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (5):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Clydebank
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Sheffield

REFERENCES:
- [Derived] Querejeta Roca G, Campbell P, Claggett B, Solomon SD, Shah AM. Right Atrial Function in Pulmonary Arterial Hypertension. Circ Cardiovasc Imaging. 2015 Nov;8(11):e003521; discussion e003521. doi: 10.1161/CIRCIMAGING.115.003521. PMID 26514759
- [Derived] Querejeta Roca G, Campbell P, Claggett B, Vazir A, Quinn D, Solomon SD, Shah AM. Impact of lowering pulmonary vascular resistance on right and left ventricular deformation in pulmonary arterial hypertension. Eur J Heart Fail. 2015 Jan;17(1):63-73. doi: 10.1002/ejhf.177. Epub 2014 Nov 4. PMID 25367310
- [Derived] Shah AM, Campbell P, Rocha GQ, Peacock A, Barst RJ, Quinn D, Solomon SD; IMPRES Investigators. Effect of imatinib as add-on therapy on echocardiographic measures of right ventricular function in patients with significant pulmonary arterial hypertension. Eur Heart J. 2015 Mar 7;36(10):623-32. doi: 10.1093/eurheartj/ehu035. Epub 2014 Feb 23. PMID 24566799
- [Derived] Hoeper MM, Barst RJ, Bourge RC, Feldman J, Frost AE, Galie N, Gomez-Sanchez MA, Grimminger F, Grunig E, Hassoun PM, Morrell NW, Peacock AJ, Satoh T, Simonneau G, Tapson VF, Torres F, Lawrence D, Quinn DA, Ghofrani HA. Imatinib mesylate as add-on therapy for pulmonary arterial hypertension: results of the randomized IMPRES study. Circulation. 2013 Mar 12;127(10):1128-38. doi: 10.1161/CIRCULATIONAHA.112.000765. Epub 2013 Feb 12. PMID 23403476
- See also: Related Info — http://www.phclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 326 participants were screened, 202 participants were randomized (103 to Imatinib and 99 to placebo). Out of 202 participants randomized 201 participants received study drug treatment (103 received imatinib mesylate, 98 received placebo). One participant was randomized to the placebo group but did not receive any study treatment.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to imatinib mesylate or placebo.
Period: Overall Study
Arm/Group | Imatinib Mesylate | Placebo
Started | 103 | 99
Completed | 69 | 81
Not Completed | 34 | 18
Not completed — Adverse Event | 27 | 7
Not completed — Lack of Efficacy | 1 | 5
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Abnormal labs | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Administration problem | 0 | 1

BASELINE CHARACTERISTICS:
Population: Age set includes all randomized participants (202). Gender set includes all treated participants (201). One participant was randomized to placebo but did not receive stuy drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate | Placebo | Total
Number analyzed (Participants) | 103 | 99 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (15.33) | 46.5 (13.60) | 48.3 (14.59)
Gender [Number; unit: participants] — One participant was randomized to placebo but did not receive study drug.
  participants
    Female | 83 | 79 | 162
    Male | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Difference in Six-minute Walk Distance Test (6MWD) Between Imatinib and Placebo at 24 Weeks
Description: This standardized walk course was 30 meters in length. During the walk the participant was connected to a portable pulse oximeter via a finger probe. Participants were instructed to walk at a comfortable speed for as far as they could manage in 6 minutes. The total distance walked (in meters) was recorded. Results were compared between the 2 groups.
Time Frame: 24 weeks
Population: The Full Analysis Set includes all participants who received at least one dose of study drug and completed the 6MWD Six-minute walk test at week 24. Repeated measurement model was used for this analysis.
Measure: Least Squares Mean (Standard Error); unit: meters
Groups:
- Imatinib: imatinib mesylate
- Placebo: Placebo to imatinib
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 92 | 93
meters | 382.94 (9.790) | 351.18 (9.834)

2. Secondary Outcome: Clinical Worsening Comparing Imatinib Versus Placebo for Adjudicated Cases
Description: Clinical worsening per participant was measured by the onset of any adjudicated event (all cause mortality; overnight hospitalization for worsening of Pulmonary Arterial Hypertension (PAH); worsening of WHO functional class by one level; 15% decline in Six Minute Walk Distance (6MWD) measured on two consecutive occasions) at 24 weeks treatment, comparing imatinib to placebo groups. A cox regression analysis model was used.
Time Frame: 24 weeks
Population: The Full Analysis Set included all participants who received at least one dose of study drug and experienced an adjudicated event. A cox regression analysis model was used.
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 37 | 32
percentage of participants | 35.9 | 32.7

3. Secondary Outcome: Change From Baseline in Right Atrial Pressure
Description: Change from baseline in right atrial pressure (mmHg) was measured via right heart catheterization according to the local hospital procedures. The right atrial pressure was assessed when the participant was in a stable hemodynamic rest state. A higher right atrial pressure number indicates worsening.
Time Frame: baseline and week 24
Population: Participants from the Full Analysis Set, defined as all randomized participants who received at least one dose of study drug, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 73 | 81
mm Hg | -1.02 (0.851) | 0.68 (0.855)

4. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure
Description: Change from baseline in mean pulmonary arterial pressure (mmHg) was measured via right heart catheterization according to the local hospital procedures. The mean pulmonary arterial pressure was assessed when the participant was in a stable hemodynamic rest state. A higher mean pulmonary arterial pressure number indicates worsening.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 75 | 82
mm Hg | -3.54 (1.585) | 1.63 (1.586)

5. Secondary Outcome: Change From Baseline in Mean Pulmonary Capillary Wedge Pressure
Description: Change from baseline in mean pulmonary capillary wedge pressure (mmHg)was measured via right heart catheterization according to the local hospital procedures. The right atrial mean pulmonary capillary wedge pressure was assessed when the participant was in a stable hemodynamic rest state.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 74 | 80
mm Hg | 0.92 (0.693) | -0.05 (0.701)

6. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance
Description: Change from baseline in systemic vascular resistance (dynes*sec*cm^-5) was measured via right heart catheterization according to the local hospital procedures. The systemic vascular resistance was assessed when the participant was in a stable hemodynamic rest state. Reduction from baseline in mean systemic vascular resistance indicates improvement.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: dynes*sec*cm^-5
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 71 | 76
dynes*sec*cm^-5 | -467.84 (78.577) | -88.10 (77.183)

7. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance
Description: Change from baseline in pulmonary vascular resistance (dynes*sec*cm^-5) was measured via right heart catheterization according to the local hospital procedures. The pulmonary vascular resistance was assessed when the participant was in a stable hemodynamic rest state. Reduction from baseline in pulmonary vascular resistance indicates improvement.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: dynes*sec*cm^-5
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 74 | 80
dynes*sec*cm^-5 | -366.47 (67.673) | 12.12 (68.963)

8. Secondary Outcome: Change From Baseline in Pulmonary Resistance Index
Description: Change from baseline in pulmonary resistance index (dynes*sec*cm^-5/m2) was measured via right heart catheterization according to the local hospital procedures. The pulmonary resistance index was assessed when the participant was in a stable hemodynamic rest state. A reduction from baseline in pulmonary resistance index indicates improvement.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: dynes*sec*cm^-5/m2
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 74 | 80
dynes*sec*cm^-5/m2 | -221.29 (47.355) | 21.92 (48.247)

9. Secondary Outcome: Change From Baseline in Cardiac Output
Description: Change from baseline in cardiac output (L/min) was measured via right heart catheterization according to the local hospital procedures. The cardiac output was assessed when the participant was in a stable hemodynamic rest state. An increase from baseline (higher number) in cardiac output indicates improvement.
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 75 | 81
Liters/minute | 1.17 (0.182) | 0.29 (0.186)

10. Secondary Outcome: Change From Baseline in Systolic Arterial Blood Pressure
Description: Change from baseline in systolic arterial blood pressure (mmHg) was measured via right heart catheterization according to the local hospital procedures. The systolic arterial blood was assessed when the participant was in a stable hemodynamic rest state.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 73 | 78
mm Hg | -2.92 (2.298) | -1.15 (2.227)

11. Secondary Outcome: Change From Baseline in Diastolic Arterial Blood Pressure
Description: Change from baseline in diastolic arterial blood pressure (mmHg) was measured via right heart catheterization according to the local hospital procedures. The diastolic arterial blood pressure was assessed when the participant was in a stable hemodynamic rest state.
Time Frame: baseline and week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 72 | 78
mm Hg | -3.81 (1.958) | -1.48 (1.909)

12. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in heart rate (bpm) was measured via right heart catheterization according to the local hospital procedures. The heart rate was assessed when the participant was in a stable hemodynamic rest state.
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 73 | 77
bpm | 0.38 (12.63) | 0.73 (2.255)

13. Secondary Outcome: Change in Borg Dyspnea Score During 6-minute Walk Test
Description: Change in Borg scale was measured at different time points at week 24. The Borg Scale consists of scale range of 0 to 10. Participants pointed to indicate their level of dyspnea before and at the end of exercise testing (where 0 indicates no breathlessness at all and 10 indicates maximum breathlessness). A reduction in this score indicates an improvement.
Time Frame: week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 92 | 91
units on a scale
  Resting (n= 86 imatinib; 89 placebo) | -0.06 (1.097) | -0.12 (1.142)
  End of test (n= 92 imatinib; 91 placebo) | -0.38 (2.009) | -0.24 (2.093)
  2 min after end (n= 82 imatinib; 81 placebo) | -0.37 (1.409) | -0.18 (1.550)
  End of test - Resting (n= 81 imatinib; 81 placebo) | -0.24 (1.193) | -0.29 (1.279)
  2 min after end - end of test (n= 82 ima; 81plb) | -0.07 (1.533) | -0.03 (1.743)

14. Secondary Outcome: Covariance of End of Study CAMPHOR Score
Description: The CAMPHOR test consists of 65 items and 3 scales. Two scales measure Health Related Quality of Life. 1) Symptoms: consists of 25 items measuring loss or abnormality of psychological, physiological or anatomical structure or function; further sub-divided into 3 subscales (energy, breathlessness and mood), 2) Disability: consists of 15 items measuring any restriction or lack of ability to perform an activity. 3) Quality of Life (QOL): consists of 25 items defining how individuals perceived ability and capacity to satisfy their needs. The 25-item symptom and QOL scales score from 0-25 where a higher score indicates the presence of more symptoms and poor QOL, respectively. The 15-item functioning scale scores 0-30; a higher score indicates poor functioning.
Time Frame: Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 45 | 44
units on a scale
  Symptoms score | 7.93 (1.372) | 9.03 (1.431)
  Activity score | 8.99 (1.177) | 10.55 (1.223)
  Quality of life score | 7.45 (1.026) | 7.13 (1.066)

15. Secondary Outcome: Plasma Concentration of QTI571 200 mg and Its Metabolite (GCP74588) Pre-dose and Between 0 Hour to 3 Hour Post-dose Per Participant
Description: Blood samples were taken from each subject participating in the study (placebo group and active treatment group) once predose and once between 0 hour to 3 hour post dose at day 1 (baseline), day 14, day 28 and day 168.
  The parent compound QTI571 and its active metabolite, GCP74588, were measured in plasma by validated liquid chromatography-mass spectrometry (HPLC-MS/MS) assay.
Time Frame: predose and between 0 hour to 3 hour post dose at day 1, day 14, day 28 and day 168
Population: The Full Analysis Set includes all patients who received at least one dose of study drug with available blood samples for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Imatinib 200 mg: imatinib mesylate 200 mg once daily
- GCP74588: imatinib metabolite
Arm/Group | Imatinib 200 mg | GCP74588
Number analyzed (Participants) | 77 | 77
ng/mL
  Day 1 - predose (n=77 imat; n=77 GCP) | 0 (0) | 0 (0)
  Day 1 - 0-3h post-dose (n=77 imat; n=77 GCP) | 471.9 (560.1) | 61.8 (77.6)
  Day 14 - predose (n=18 imat; n=18 GCP) | 579.6 (384.9) | 178.8 (122.8)
  Day 14 - 0-3h post-dose (n=19 imat; n=19 GCP) | 1005.7 (665.6) | 233.8 (170.9)
  Day 28 - predose (n=20 imat; n=20 GCP) | 658.8 (450.3) | 228.6 (121.4)
  Day 28 - 0-3h post-dose (n=19 imat; n=19 GCP) | 1438.6 (924.4) | 323.9 (150.6)
  Day 168 predose (n=24 imat; n=24 GCP) | 398.6 (415.5) | 126.6 (83.3)
  Day 168- 0-3h post-dose (n=23 imat; n=23 GCP) | 710.8 (639.7) | 166.1 (103.1)

16. Secondary Outcome: Plasma Concentration of QTI571 400 mg and Its Metabolite (GCP74588) Pre-dose and Between 0 Hour to 3 Hour Post-dose Per Participant
Description: as for outcome 15
Time Frame: predose and between 0 hour to 3 hour post dose at day 1, day 14, day 28 and day 168
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Imatinib 400 mg: imatinib mesylate 400 mg once daily
Arm/Group | Imatinib 400 mg | GCP74588
Number analyzed (Participants) | 62 | 62
ng/mL
  Day 1 - predose (n=12 imat; n=12 GCP) | 0 (0) | 0 (0)
  Day 1 - 0-3h post-dose (n=13 imat; n=13 GCP) | 843.2 (788.9) | 109.9 (132.4)
  Day 14 - predose (n=62 imat; n=62 GCP) | 516.5 (405.2) | 155.1 (101.1)
  Day 14 - 0-3h post-dose (n=62 imat; n=62 GCP) | 1172.8 (1088.9) | 233.7 (165.6)
  Day 28 - predose (n=55 imat; n=55 GCP) | 829.8 (482.6) | 248.2 (125.2)
  Day 28 - 0-3h post-dose (n=58 imat; n=58 GCP) | 1335.3 (817.9) | 320.7 (154.8)
  Day 168 predose (n=36 imat; n=36 GCP) | 869.9 (407.8) | 241.4 (91.9)
  Day 168- 0-3h post-dose (n=35 imat; n=35 GCP) | 1616.1 (787.6) | 348.0 (119.1)

ADVERSE EVENTS:
Description: 202 participants were randomized (103 imatinib & 99 placebo; however, one participant who was randomized to the placebo group did not receive study drug and was excluded from this analysis set. The safety set includes all participants who received study drug = 201 (103 imatinib, 98 placebo).
Arm/Group | Imatinib | Placebo
Serious Adverse Events (participants affected / at risk) | 45/103 | 29/98
Other Adverse Events (participants affected / at risk) | 96/103 | 80/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=103) | Placebo (N=98)
Anaemia (Blood and lymphatic system disorders) | 7 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 2
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Device leakage (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection site extravasation (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 6 | 0
Pyrexia (General disorders) | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 3 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Cardiac output decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Right atrial pressure increased (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 5 | 0
Syncope (Nervous system disorders) | 1 | 5
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypoperfusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=103) | Placebo (N=98)
Anaemia (Blood and lymphatic system disorders) | 8 | 2
Palpitations (Cardiac disorders) | 4 | 7
Periorbital oedema (Eye disorders) | 30 | 7
Abdominal distension (Gastrointestinal disorders) | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 33 | 18
Dyspepsia (Gastrointestinal disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 56 | 23
Vomiting (Gastrointestinal disorders) | 30 | 10
Face oedema (General disorders) | 9 | 1
Fatigue (General disorders) | 10 | 7
Non-cardiac chest pain (General disorders) | 3 | 5
Oedema peripheral (General disorders) | 41 | 20
Pyrexia (General disorders) | 7 | 3
Device related infection (Infections and infestations) | 1 | 5
Influenza (Infections and infestations) | 2 | 5
Nasopharyngitis (Infections and infestations) | 18 | 19
Respiratory tract infection (Infections and infestations) | 3 | 7
Sinusitis (Infections and infestations) | 2 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 7
Urinary tract infection (Infections and infestations) | 4 | 5
Blood creatinine increased (Investigations) | 9 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Dizziness (Nervous system disorders) | 8 | 5
Headache (Nervous system disorders) | 25 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.